CLINICAL TRIAL: NCT02789579
Title: The Preventive Urinary Tract Infection Role of One Week Solutions of Antimicrobial Application Before Minimally Invasive Upper Tract Lithotomy
Brief Title: The Preventive Infection Role of One Week Antibiotics Before Minimally Invasive Upper Tract Lithotomy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: XH-16-010
Record Dates: First submitted 2016-04-15; First posted 2016-06-03 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Complication of Surgical Procedure
Keywords: prophylactic; Urinary Tract Infections; Minimally invasive upper tract lithotomy
MeSH Terms: conditions — Urinary Tract Infections | interventions — Levofloxacin; Nitrofurantoin; Cefuroxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- levofloxacin 3 days group (Experimental): There are 30 patients in the group,each patient meets the eligibility criteria and does not meet the exclusion criteria,and receives levofloxacin 0.5g,qd,po 3 days before Minimally invasive upper tract lithotomy.
  Interventions: Drug: levofloxacin; Drug: cefuroxime
- nitrofurantoin 3 days group (Experimental): There are 30 patients in the group,each patient meets the eligibility criteria and does not meet the exclusion criteria,and receives nitrofurantoin 0.1g, tid, po 3 days before Minimally invasive upper tract lithotomy.
  Interventions: Drug: Nitrofurantoin; Drug: cefuroxime
- cefuroxime group (Experimental): There are 150 patients in the group,each patient meets the eligibility criteria and does not meet the exclusion criteria,and does not receive oral antibiotics 7 days before Minimally invasive upper tract lithotomy.All patients in all groups, 30 minutes before surgery, are given preventive medication cefuroxime 1.5g ivgtt, and continue using 1.5g q12h ivgtt until postoperative 48 hours.
  Interventions: Drug: cefuroxime
- levofloxacin 7 days group (Experimental): There are 30 patients in the group,each patient meets the eligibility criteria and does not meet the exclusion criteria,and receives levofloxacin 0.5g,qd,po 7 days before Minimally invasive upper tract lithotomy.
  Interventions: Drug: levofloxacin; Drug: cefuroxime
- nitrofurantoin 7 days group (Experimental): There are 30 patients in the group,each patient meets the eligibility criteria and does not meet the exclusion criteria,and receives nitrofurantoin 0.1g, tid, po 7 days before Minimally invasive upper tract lithotomy.
  Interventions: Drug: Nitrofurantoin; Drug: cefuroxime

INTERVENTIONS:
Drug: levofloxacin — There are 50 patients in the group,each patient receives levofloxacin 0.5g, qd, po 7 days before Minimally invasive upper tract lithotomy.All patients in all groups, 30 minutes before surgery, are given preventive medication cefuroxime 1.5g ivgtt, and continue using 1.5g q12h ivgtt until postoperative 48 hours.
  Other Names: Cravit
  Arms: levofloxacin 3 days group; levofloxacin 7 days group
Drug: Nitrofurantoin — There are 50 patients in the group,each patient receives nitrofurantoin 0.1g, qd, po 7 days before Minimally invasive upper tract lithotomy.All patients in all groups, 30 minutes before surgery, are given preventive medication cefuroxime 1.5g ivgtt, and continue using 1.5g q12h ivgtt until postoperative 48 hours.
  Other Names: Furadantin
  Arms: nitrofurantoin 3 days group; nitrofurantoin 7 days group
Drug: cefuroxime — There are 150 patients in the group, 30 minutes before surgery, each patient is given preventive medication cefuroxime 1.5g ivgtt, and continue using 1.5g q12h ivgtt until postoperative 48 hours.
  Other Names: zinacef

SUMMARY:
Minimally invasive upper tract lithotomy is currently a common operation method on treatment of urinary tract stones, but the postoperative complication urinary tract infection or urinary sepsis has turned into a serious threat to the patient's life, when severe, can result in a higher death rate.Although more the more importance were attached to, an effective prevention measures still have not been found.

Among Urinary calculi, the higher rates of infection stone resulted in a higher incidence of postoperative urinary tract infection. The conventional postoperative prophylaxis medicine was the use of antimicrobial drugs half an hour before surgery.Foreign studies had shown that continuous preoperative one week use of nitrofurantoin can significantly reduce the incidence of urinary sepsis. So the investigators assume that preoperative extended use time of prophylaxis antibiotic may reduce the incidence of urinary tract infection or urinary sepsis.

This study uses a computerized random method. According to preoperative use of different antimicrobial drug or treatment, all patients are randomly divided into five groups, namely levofloxacin 3days group,levofloxacin 7days group, nitrofurantoin 3days group,nitrofurantoin 7days group and cefuroxime group.The levofloxacin group receives levofloxacin 0.5g, qd, po, the nitrofurantoin group was given oral nitrofurantoin 100mg, tid, po.to explore the better antibiotics types, medication timing and duration of treatment to prevent postoperative infection after minimally invasive upper tract lithotomy, so as to reduce the incidence of postoperative urinary tract infection or sepsis.

DETAILED DESCRIPTION:
1. Sample Calculation: Based on the literature, the occurrence rate of fever after Percutaneous Nephrolithotripsy (PCNL) was 21% -39.8%, urinary tract infection rate 38%, SIRS rate 11.2%, the incidence rate of urinary sepsis 0.3% - 4.7%,and the mortality rate with sepsis was 60% -80%. Expected incidence rate of urinary tract infection decreased to 23%, and the difference is statistically significant. Provided that the case of the two groups is equal, the expected strength of evidence is 0.9, α = 0.05, the lost up to 20%, the investigators calculated that the minimum sample size required is 150 cases. Urology department has 70 ward beds with PCNL surgery or Flexible Ureteroscopy Lithotripsy (FURL) about 400 cases per year, and the sample size can meet the study requirements. All cases are from outpatient or emergency department.
2. Grouping and medication: This study uses a computerized random method. According to preoperative use of different antimicrobial drug or treatment, all patients are randomly divided into five groups, namely levofloxacin 3days group,levofloxacin 7days group, nitrofurantoin 3days group,nitrofurantoin 7days group and cefuroxime group.and each group of levofloxacin group or nitrofurantoin group has been given prophylactic for 3 or 7 days. The levofloxacin group receives levofloxacin 0.5g, qd, po, the nitrofurantoin group was given oral nitrofurantoin 100mg, tid, po. All patients in cefuroxime group, 30 minutes before surgery, are given preventive medication cefuroxime 1.5g ivgtt, and continue using 1.5g q12h ivgtt until postoperative 48 hours.
3. Sterilization or bacterial culture: Surgical areas is disinfected with 10% povidone-iodine, all surgical instruments are sterilized by high-temperature steam. after renal pelvises are punctured, some urine is extracted for bacterial culture. Stones removed by surgery are fragmented into small fragments, and stored at 36.5 ℃ tubes within a day in order to facilitate the proliferation of bacteria, then grown in culture medium for bacterial culture.
4. Preoperative items observed: urinalysis, urine culture, renal function, blood, CRP, procalcitonin, bacterial endotoxin test, kidney function, body temperature changes prophylactic or preoperative. Imaging tests include urinary tract calculi line pyelography and CT.
5. Postoperative follow-up: urine, urine culture, renal function, blood routine, CRP, procalcitonin, bacterial endotoxin test, renal function and urinary tract stones line urography and CT examination were made in all patients. Vital signs such as body temperature, heart rate and blood pressure once every two hours were monitored in 48 hours, and were monitored every 4 hours after 48 hours. Blood routine was checked daily until 3 days postoperative or 48 hours after abatement of fever. When white blood cell count> 12 × 109 / L and / or body temperature> 38 ℃ °, it is considered to be systemic inflammatory response (SIRS, modified Sepsis Diagnostic Criteria). Renal fistula was retained for 48 hours Postoperative, and pleural effusion fistula was removed if there was no fever after it was pinched 24 hours.
6. Statistical analysis: Statistical Product and Service Solutions (SPSS)19.0 statistical software was used for analysis. Count data were analyzed by analysis of variance or t Test. Measurement data were analyzed by Chi-square Test. The results were evaluated within the safe range of 95%,when P <0.05,it was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of urinary tract lithiasis (stones ≥ 2cm) or urolithiasis with hydronephrosis

Exclusion Criteria:

* antimicrobial drugs been administered in the latest month
* immunosuppressor been administered in the latest month
* urinary tract infection or positive urine culture results
* history of urinary calculi surgery
* diabetes
* chronic renal failure patients
* neurogenic bladder dysfunction
* abnormal anatomy of the kidney
* neuromuscular dysfunction (spina bifida, paraplegia, green Barry syndrome, or quadriplegia)
* more than 90 minutes operation time
* more than 1000 ml blood loss

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically urinary tract infection confirmed by laboratory examination or urine bacterial culture. | 3 or 7 days after operation
  Compared with control group, the positive rate of operative blood routine, CRP, urine routine, urine culture, procalcitonin , bacterial endotoxin test of experimental group are declining.

SECONDARY OUTCOMES:
Evidence of clinically urosepsis confirmed by laboratory examination, urine bacterial culture, and vital signs | 3 or 7 days after operation
  Compared with control group, the positive rate of operative blood culture, procalcitonin are declining.

CONTACTS AND LOCATIONS:
Overall Officials: li lixia, Master, Principal Investigator — Xinhua Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Department of Pharmacy, Xinhua Hospital, Shanghai Jiaotong University School of Medicine.Kongjiang Road 1665,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sofikerim M, Gulmez I, Karacagil M. One week of ciprofloxacin before percutaneous nephrolithotomy significantly reduces upper tract infection and urosepsis: a prospective controlled study. BJU Int. 2007 Feb;99(2):466. doi: 10.1111/j.1464-410X.2007.06746_6.x. No abstract available. PMID 17313438
- [Result] Bag S, Kumar S, Taneja N, Sharma V, Mandal AK, Singh SK. One week of nitrofurantoin before percutaneous nephrolithotomy significantly reduces upper tract infection and urosepsis: a prospective controlled study. Urology. 2011 Jan;77(1):45-9. doi: 10.1016/j.urology.2010.03.025. Epub 2010 Jun 8. PMID 20570319